CLINICAL TRIAL: NCT02034708
Title: Intra-individual Cross-over Efficacy Evaluation of Dotarem®-Enhanced MRI Compared to Gadovist®/ Gadavist®-Enhanced MRI in the Diagnosis of Brain Tumors
Brief Title: Efficacy Evaluation of Dotarem®-Enhanced MRI Compared to Gadovist®/Gadavist®-Enhanced MRI in the Diagnosis of Brain Tumors
Acronym: REMIND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: DGD-44-058
Record Dates: First submitted 2014-01-10; First posted 2014-01-13 (Estimated); Results first posted 2016-10-25 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-11

CONDITIONS: Primary Brain Tumor
Keywords: Primary brain tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — gadoterate meglumine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dotarem®/Gadovist® (Experimental): Dotarem®-enhanced MRI, then Gadovist®/Gadavist®-enhanced MRI
  Interventions: Drug: Dotarem®; Drug: Gadovist®/Gadavist®
- Gadovist®/Dotarem® (Experimental): Gadovist®/Gadavist®-enhanced MRI then Dotarem® enhanced MRI
  Interventions: Drug: Dotarem®; Drug: Gadovist®/Gadavist®

INTERVENTIONS:
Drug: Dotarem® — Dotarem® 0.1 mmoL/kg (0.2 mL/kg), intravenous (I.V.) bolus.
Drug: Gadovist®/Gadavist® — Gadovist®/Gadavist®, 0.1mmol/kg (0.1mL/kg), intravenous (I.V.) bolus.

SUMMARY:
The purpose of this study is to demonstrate non-inferiority of Dotarem®-enhanced MRI as compared to Gadovist®/ Gadavist®-enhanced MRI in the diagnosis of brain tumors in terms of overall lesion visualization and characterization (off-site assessment).

270 patients will be randomized between 2 arms defining the sequence of administration of the contrast agents at the dose of 0.1mmol/kg, with a minimum of 48 hours and a maximum of 14 days in between.

Each patient will, therefore, receive two MRI during his/her participation in the study.

The two arms consist in :

* Dotarem® in the first MRI, then Gadovist®/Gadavist® in the second MRI.
* Gadovist®/Gadavist® in the first MRI, then Dotarem® in the second MRI.

Contrast-enhanced MRIs will be performed on 1.5 or 3 Tesla systems.

MRI examinations will be evaluated centrally by blinded independent readers for the main evaluation criterion.

ELIGIBILITY:
Inclusion Criteria:

* Female or male adult patient (patient having reached legal majority age)
* Patient with known or highly suspected primary intracranial tumors (intra-axial or extra-axial) detected by previous CT or MRI examination who are scheduled to undergo a routine contrast-enhanced MRI
* Female patient must have effective contraception throughout the study and must have a negative urine pregnancy test at inclusion, or be surgically sterilized, or post-menopausal (minimum 12 months of amenorrhea)
* Patient having provided his/her written informed consent to participate in the trial prior to any study-related procedure being conducted
* Patient with national health insurance (according to local regulatory requirements)

Exclusion Criteria:

* Patient with rapidly evolving brain tumor that could change in appearance between the time of the two study MRI examinations.
* Patient undergoing current or recent treatment within past 6 weeks or scheduled for any treatment that could results in changes of lesion appearance between the two study examinations. This would include, but not restricted to, the following: current or recent radiation therapy, surgery, starting or recent chemotherapy.
* Patient with a contraindication to MRI (e.g., pacemaker, aneurysm clip, severe claustrophobia, infusion pumps, cochlear implants metallic or others according to the imaging site standard practice)
* Patient with known severely impaired renal function (defined as eGFR MDRD< 30 ml/min/1.73m2)
* Patient with known Class III/IV congestive heart failure according to the New York Heart Association classification
* Patient with known severe adverse drug reaction or contraindication to Gadolinium-Based Contrast Agent
* Patient having received any contrast agent within 48 hours prior to first study contrast agent injection scheduled for the study and patient expected to receive any other contrast agent within 24 hours of the last study contrast agent injection
* Patient presenting with any condition which, based on the investigator's clinical judgment, would prevent the patient from completing all trial assessments and visits
* Patient under guardianship and/or unable or unwilling to cooperate with the requirements of this trial
* Pregnant or breast feeding female patient
* Patient already included in this trial
* Patient included in another clinical trial involving an IMP within 30 days before the first investigational contrast agent injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Maravilla, MD, Study Chair — University of Washington Medical Center, Seattle, USA
Locations (32):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona Medical Center, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - University of Michigan Health System, Ann Arbor, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Washington University, St Louis, Missouri
  - Winthrop University Hospital Clinical Trials Center, Mineola, New York
  - Temple University Hospital, Philadelphia, Pennsylvania
  - MUSC (Medical University of South Carolina), Charleston, South Carolina
  - UVM MRI Center for Biomedical Imaging, Burlington, Vermont
  - University of Washington Medical Center, Seattle, Washington
- Colombia (6):
  - Fundacion Abood Shaio, Bogotá
  - Fundacion Cardioinfantil Instituto de Cardiologia, Bogotá
  - Instituto Nacional de Cancerologia, Bogotá
  - Centro Medico Imbanaco, Cali
  - Fundacion Instituto de Alta Tecnologia Medica de Antioquia IATM, Medellín
  - Hospital Pablo Tobon Uribe, Medellín
- Mexico (7):
  - Hospital CIMA, Chihuahua City, Chihuahua
  - Morales Vargas Centro de Investigación S.C., León, Guanajuato
  - Centro Neurologico ABC, México, Mexico Distrito Federal
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Winsett Rethman S.A. de C.V., Monterrey, Nuevo León
  - Centro Regiomontano de Investigacion S.C., Monterrey
  - Clinical Research Institute S.C., Tlanepantla
- South Korea (5):
  - Chonbuk national Univ Hosp, Jeonju, Jeollabuk-do
  - Chungbuk National University, Cheongju-si, North Chungcheong
  - Seoul St.Mary Hospital, Seoul, Seocho-gu
  - Asan medical center, Seoul, Songpa-Gu
  - Ajou University Hospital, Suwon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients with known or highly suspected primary intracranial tumors and scheduled for a Dotarem®-enhanced MRI were recruited in 27 active centers in 4 countries (Colombia, South Korea, Mexico and United States) from June 2014 to September 2015.
Pre-assignment Details: 279 patients signed an informed consent for the study and therefore were considered as included. From these 279 patients, 11 did not receive any injection : 4 for consent withdrawn, 3 for deviation from plan specified in the protocol, 2 for adverse events, 1 at the investigator's discretion and 1 for other reason.
Groups:
- Dotarem®/Gadovist®: Dotarem®-enhanced MRI, then Gadovist®/Gadavist®-enhanced MRI
  Dotarem®: 0.1 mmoL/kg (0.2 mL/kg), intravenous (I.V.) bolus.
  Gadovist®/Gadavist®: 0.1mmol/kg (0.1mL/kg), intravenous (I.V.) bolus.
- Gadovist®/Dotarem®: Gadovist®/Gadavist®-enhanced MRI then Dotarem® enhanced MRI
  Dotarem®: 0.1 mmoL/kg (0.2 mL/kg), intravenous (I.V.) bolus.
  Gadovist®/Gadavist®: 0.1mmol/kg (0.1mL/kg), intravenous (I.V.) bolus.
Period: First Contrast Agent Injection (1 Day)
Arm/Group | Dotarem®/Gadovist® | Gadovist®/Dotarem®
Started | 138 | 130
Completed | 138 | 130
Not Completed | 0 | 0
Period: Wash-out (From 2 Days up to 14 Days)
Arm/Group | Dotarem®/Gadovist® | Gadovist®/Dotarem®
Started | 138 | 130
Completed | 129 | 120
Not Completed | 9 | 10
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 3 | 3
Not completed — other reason | 3 | 2
Period: Second Contrast Agent Injection (1 Day)
Arm/Group | Dotarem®/Gadovist® | Gadovist®/Dotarem®
Started | 129 | 120
Completed | 129 | 120
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients receiving at least one injection of contrast agent and with one valid assessment of the primary outcome
Groups:
- Total: Total of all reporting groups
Arm/Group | Dotarem®/Gadovist® | Gadovist®/Dotarem® | Total
Number analyzed (Participants) | 138 | 130 | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (15.2) | 54.4 (15.1) | 53.6 (15.1)
Gender [Count of Participants; unit: Participants]
  Female | 87 | 85 | 172
  Male | 51 | 45 | 96
Region of Enrollment [Number; unit: participants]
  Colombia | 16 | 16 | 32
  United States | 46 | 40 | 86
  Korea, Republic of | 24 | 23 | 47
  Mexico | 52 | 51 | 103
Body Mass Index [Mean (Standard Deviation); unit: kg per square metre] | 27.71 (5.35) | 27.62 (5.23) | 27.66 (5.28)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Overall Lesion Visualization and Characterization Scored as Good or Excellent
Description: Overall lesion visualization and characterization, based on assessment of the primary or largest lesion if there is more than one lesion present, was assessed by 3 independent off-site readers on a 4-point scale:
  0. Poor: does not allow adequate visualization and characterization of the lesion; 1. Fair: allows partial visualization and characterization of the lesion ; 2. Good: allows adequate visualization and characterization of the lesion; 3. Excellent: allows excellent visualization and characterization of the lesion.
Time Frame: Up to 15 days after randomization
Population: Patients with at least one valid assessment of the primary outcome and without major protocol deviation
Measure: Number; unit: percentage of patients
Groups:
- Gadovist® (Reader 1): Patients who received Gadovist® Results for reader 1
- Dotarem® (Reader 1): Patients who received Dotarem® Results for reader 1
- Gadovist® (Reader 2): Patients who received Gadovist® Results for reader 2
- Dotarem® (Reader 2): Patients who received Dotarem® Results for reader 2
- Gadovist® (Reader 3): Patients who received Gadovist® Results for reader 3
- Dotarem® (Reader 3): Patients who received Dotarem® Results for reader 3
Arm/Group | Gadovist® (Reader 1) | Dotarem® (Reader 1) | Gadovist® (Reader 2) | Dotarem® (Reader 2) | Gadovist® (Reader 3) | Dotarem® (Reader 3)
Number analyzed (Participants) | 234 | 234 | 234 | 234 | 234 | 234
percentage of patients | 94.0 | 96.2 | 93.2 | 90.6 | 99.6 | 100.0

ADVERSE EVENTS:
Time Frame: From patient inclusion up to 30 min after last contrast agent injection
Groups:
- Dotarem®: Patients who received Dotarem®
- Gadovist®: Patients who received Gadovist®
- Total: Patients who received at least one injection of contrast agent
Arm/Group | Dotarem® | Gadovist® | Total
Serious Adverse Events (participants affected / at risk) | 1/258 | 0/259 | 1/268
Other Adverse Events (participants affected / at risk) | 42/258 | 44/259 | 63/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dotarem® (N=258) | Gadovist® (N=259) | Total (N=268)
Aggravation of existing disorder (General disorders) | 1 (1) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dotarem® (N=258) | Gadovist® (N=259) | Total (N=268)
Injection site pain (General disorders) | 12 (12) | 12 (13) | 20 (25)
Medical device pain (General disorders) | 15 (15) | 17 (17) | 17 (32)
Injection site coldness (General disorders) | 1 (1) | 1 (1) | 2 (2)
Injection site paraesthesia (General disorders) | 2 (2) | 1 (1) | 2 (3)
Catheter site related reaction (General disorders) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Drug ineffective (General disorders) | 0 (0) | 1 (1) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site inflammation (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 4 (4) | 3 (3) | 7 (7)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4) | 5 (6)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 5 (5)
Infrequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each investigator agrees not to publish/present the results of the study main criterion involving only the patients included in his/her center. Publications on specific topics can be performed only after main publication.The sponsor can review the publication at least 30 days before the submission to the scientific review and any abstract project at least 10 working days before submission to the congress scientific committee. The sponsor can require changes to the publication or the abstract.